CLINICAL TRIAL: NCT02210351
Title: Evaluation of Association Between Apical Dysfunction and Trans Apical Access for TAVR, in Patients With Severe Aortic Stenosis, Undergoing Trans Apical Trans Catheter Aortic Valve Replacement (TAP-TAVR).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Danny Spiegelstein, Dr. Danny Spiegelstein, Physician, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-13-0829-DS-CTIL
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Severe Symptomatic Aortic Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI test (Experimental)
  Interventions: Device: MRI test

INTERVENTIONS:
Device: MRI test

SUMMARY:
The asses and evaluate whether trans apical access for TAVR is associated with apical dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis defined as aortic valve area of less than 1 cm2 or index area of 0.6 cm2/m2 by echocardiography.
2. Symptomatic patients with aortic stenosis referred for medically indicated AVR
3. Signed informed consent to participate in the study.

Exclusion Criteria:

1. Inability to sign written informed consent.
2. Abnormal Apical dysfunction at baseline
3. LVEF < 20%
4. Pregnancy or breast feeding.
5. Need for emergency surgery for any reason.
6. Any case in which the practicing physician asserts that enrollment in the protocol will

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricle ejection fraction | two months after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Leviev Heart Center, Sheba Medical Center, Ramat Gan, Israel